CLINICAL TRIAL: NCT02805751
Title: Mechanical Properties in Conservative Treated Achilles Tendon Ruptures With or Without Early Controlled Loading
Brief Title: Early Controlled Loading on Conservative Treated Achilles Tendon Ruptures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Pernilla Eliasson, Postdoc, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Early loading
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2016-06

CONDITIONS: Tendon Injuries; Soft Tissue Injuries; Achilles Tendon Rupture
Keywords: Achilles; Tendon; Loading; Rehabilitation
MeSH Terms: conditions — Tendon Injuries; Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): This constitutes the currently accepted regime and is therefore consider the control group (CTRL) with early range of motion and early weight bearing. The control group was allowed to have weight-bearing as tolerated from day 0. They are also instructed to perform tendon strain exercises 3 times each day from 2 weeks after the rupture.
  Interventions: Other: Tendon strain exercises; Other: Early weight bearing
- Early loading (Experimental): The patients in the early loading group are also allowed to have weight-bearing as tolerated from day 0 and perform tendon strain exercises 3 times each day from 2 weeks after the rupture. The patients in this group will also remove the walker twice a day and use a special training pedal for 5 weeks (until walker removal).
  Interventions: Device: Early loading on a training pedal; Other: Tendon strain exercises; Other: Early weight bearing

INTERVENTIONS:
Device: Early loading on a training pedal — The patients will perform early loading by using a special training pedal for 5 weeks, starting 2 weeks after the rupture. The patients will remove the walker and train twice a day on this pedal.
  Arms: Early loading
Other: Tendon strain exercises — The patients will perform tendon strain exercises 3 times each day from 2 weeks after the rupture.
Other: Early weight bearing — The patients are allowed to bear weight as much as tolerated in the walker from day 1.

SUMMARY:
The purpose of this study is to measure the mechanical properties of the tendon after conservative treated Achilles tendon ruptures with or without early controlled loading. This is done in a randomized trial and the mechanical properties are measured using roentgen stereometric analysis (RSA).

The hypothesis is that early weightbearing improves mechanical properties of conservative treated Achilles tendon ruptures without causing elongation of the tendon.

DETAILED DESCRIPTION:
Treatment of Achilles tendon ruptures includes surgical repair or immobilization in an orthosis, followed by prolonged rehabilitation. Improved rehabilitation regimens still display imperfect recovery, with deficits such as persistent end-range muscle weakness, tendon elongation and incomplete return to pre-injury activity level. The underlying mechanisms are unknown, but are likely to involve molecular and cellular aspects of the early healing processes. Animal experiments have shown that short episodes of vigorous loading during tendon healing create a stronger tendon, and lead to less elongation than continuous loading. Early controlled training has also been shown to improve the material properties of surgically repaired tendons. However, more and more clinics now turn away from surgery and towards conservative treatment, while studies on rehabilitation mainly concern sutured tendons. It is therefore also important to understand how to best rehabilitate conservatively treated patients. The aim is to investigate the effect of early controlled loading on conservatively treated Achilles tendon ruptures.

The patients (age 18-60 years of age) are treated conservatively by receiving a removable foam walker boot at the emergency department. The patients are thereafter called by the principal investigator and are asked if they want to participate in the study. Patients who are interested in participating in the study receive oral and in written information about the study of the principal investigator of the study (Pernilla Eliasson).

After 2 weeks, the rupture is localized by ultrasound and 4 tantalum beads are implanted percutaneously in the proximal and distal part of the tendon. These beads are used for measurements of the mechanical properties of the tendon by using RSA.

The patients are thereafter randomized to early controlled loading or control.

All patients wear the foam walker boot for 7 weeks. Full weight-bearing is allowed as tolerated from the beginning. Both groups perform motion exercises outside the boot with 20 repetitions, 3 times per day as of 14 days after rupture.

The patients in the early loading group are provided with a special training pedal where pedal resistance can be increased during the treatment period. The patients will use this pedal twice a day starting 2 weeks after rupture.

After the initial 7 weeks, the patients are referred to physical therapists uninvolved in this research, but with the instruction to follow the regional rehabilitation guidelines for Achilles tendon ruptures.

Mechanical properties of the tendon will be estimated by measuring tendon length, cross-sectional area (CSA) and stiffness at week 7, 19 and 52.

The elastic modulus of the tendon at 19 weeks it the primary variable of this study.

At week 7, both the elastic and plastic deformation will be measured. Tendon CSA will be evaluated using computer tomography (CT). Tendon elongation will be evaluated by RSA at week 2, 7, 19 and 52. Calf muscle circumference, passive and active range of motion in the ankle joint and a heel-raise test will be performed at week 19 and 52.

The overall function will be assessed by the Achilles Tendon Rupture Score at 19 and 52 weeks.

Complications and re-ruptures will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Complete Achilles tendon rupture placed in the mid-substance of the Achilles tendon
* Presented within 14 days from injury
* 18-60 years old

Exclusion Criteria:

* Inability to understand swedish
* previous injured tendon
* Diabetes mellitus
* History of Rheumatoid disease
* Treatment with steroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Modulus of Elasticity | 19 weeks
  Modulus of elasticity will be measured using RSA and measurements of the distance between tantalum beads. A certain frame is used allowing us to apply a pedal to the forefoot and load it with weights. Tendon size will be measured using CT.

SECONDARY OUTCOMES:
Tendon elongation | 2, 7, 19 and 52 weeks after rupture
  Tendon elongation will be evaluated using RSA and measurements of the distance between tantalum beads
Modulus of Elasticity | 7 and 52 weeks after rupture
  Modulus of elasticity will be measured using RSA and measurements of the distance between tantalum beads. A certain frame is used allowing us to apply a pedal to the forefoot and load it with weights. Tendon size will be measured using CT.
Achilles tendon total rupture score (ATRS) | 19 and 52 weeks after rupture
  Patient reported outcome regarding function in their Achilles tendon
Maximal range of motion | 19 and 52 weeks after rupture
  The maximun range of motion in the ankle joint will be measured in plantar and dorsiflexion.
Heel-rise | 19 and 52 weeks after rupture
  The number of heel-rises and the heel-rise height will be used for calculation of the heel-rise work.
Plastic deformation of the tendon | 7 weeks after rupture
  Plastic deformation will be measured using RSA and measurements of the distance between tantalum beads while the patient continues to have a load on the tendon for 3 minutes with a weight. Tendon size will be measured using CT.
Calf muscle circumference | 19 and 52 weeks
  Measurement of the circumference at the thickest part of the calf

CONTACTS AND LOCATIONS:
Overall Officials: Per Aspenberg, MD, PhD, Study Director — Linkoeping University
Locations (1):
- University Hospital Linkoeping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rendek Z, Bon Beckman L, Schepull T, Danmark I, Aspenberg P, Schilcher J, Eliasson P. Early Tensile Loading in Nonsurgically Treated Achilles Tendon Ruptures Leads to a Larger Tendon Callus and a Lower Elastic Modulus: A Randomized Controlled Trial. Am J Sports Med. 2022 Oct;50(12):3286-3298. doi: 10.1177/03635465221117780. Epub 2022 Aug 25. PMID 36005394